CLINICAL TRIAL: NCT06855524
Title: Fucoidan for Patients With Chemotherapy-Related Fatigue: A Double-Blind, Randomized, Placebo-Controlled Pilot Study
Brief Title: Fucoidan for Preventing Chemotherapy-Related Fatigue in Patients With Gastrointestinal or Gynecological Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: MC231007; NCI-2025-01334 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-004592 (Other: Mayo Clinic Institutional Review Board); MC231007 (Other: Mayo Clinic)
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Malignant Digestive System Neoplasm; Malignant Female Reproductive System Neoplasm
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Research staff, other than pharmacy, are blinded and will dispense the fucoidan or placebo to the patient at the site.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (fucoidan) (Experimental): Patients receive fucoidan PO TID for 8 weeks. After completion of fucoidan, patients then cross over into Arm 2 for 8 weeks. Patients may optionally undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Dietary Supplement: Oligo-fucoidan; Other: Questionnaire Administration
- Arm 2 (placebo) (Placebo Comparator): Patients receive placebo PO TID for 8 weeks. After completion of placebo, patients then cross over into Arm 1 for 8 weeks. Patients may optionally undergo blood sample collection during screening and on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Dietary Supplement: Oligo-fucoidan — Given PO
  Other Names: Low-molecular-weight Fucoidan; Oligo Fucoidan
  Arms: Arm 1 (fucoidan)
Drug: Placebo Administration — Given PO
  Arms: Arm 2 (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests how well fucoidan works in preventing chemotherapy-related fatigue compared to a placebo in patients with gastrointestinal (GI) or gynecological (GYN) cancer. Fatigue poses a burden in patients with malignancies undergoing systemic chemotherapy. Fucoidan is a dietary supplement made of complex sugar that contain sulfate groups attached to their sugar units (sulfated polysaccharide) which found in brown seaweed. It is thought to have anti-inflammatory, anti-viral, anti-thrombotic, anti-diabetic, and anti-tumor effects in pre-clinical models. Giving fucoidan may be effective in preventing chemotherapy-related fatigue in patients with GI or GYN.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of fucoidan versus (vs.) placebo in preventing fatigue as assessed by a single-item measure of fatigue at 8 weeks following the initiation of platinum-based doublet/triplet.

SECONDARY OBJECTIVES:

I. To estimate 1) changes in fatigue via the single item measure of fatigue from baseline to week 16 2) the Global Impression of Change at week 8 and week 16 and 3) the Functional Assessment of Cancer Therapy-Fatigue (FACT-F) subscale at week 8 and week 16.

II. To evaluate the frequency and severity of toxicity as reported by the patient on the Symptom Experience Diary.

EXPLORATORY OBJECTIVE:

I. To evaluate if there are differences in inflammatory markers C-reactive protein (CRP) and IL-6 between groups from baseline to week 8.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM 1: Patients receive fucoidan orally (PO) three times a day (TID) for 8 weeks. After completion of fucoidan, patients then cross over into Arm 2 for 8 weeks. Patients may optionally undergo blood sample collection during screening and on study.

ARM 2: Patients receive placebo PO TID for 8 weeks. After completion of placebo, patients then cross over into Arm 1 for 8 weeks. Patients may optionally undergo blood sample collection during screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance score 0 or 1
* Starting platinum-based doublet/triplet therapy for gynecologic or gastrointestinal cancer in the non-curative setting, with at least 16 weeks of chemotherapy and/or immunotherapy planned prior to registration; able to start study treatment ≤ 7 days prior to starting chemotherapy
* Life expectancy at least 6 months
* Hemoglobin ≥ 10 g/dL (obtained ≤ 30 days prior to registration)
* Creatinine ≤ 1.5 x upper normal limit (UNL) OR calculated creatinine clearance ≥ 50 ml/min using the Cockcroft-Gault (obtained ≤ 30 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 1.5 x UNL; [≤ 5 x upper limit of normal (ULN) for patients with liver involvement] (obtained ≤ 30 days prior to registration)
* Ability to complete patient questionnaires alone or with assistance and to be willing to be contacted by study staff
* Provide written informed consent
* Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Willing to use a highly effective method of contraception from the first dose of study medication through 30 days after the last dose of study medication, for persons of childbearing potential or persons able to father a child only
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study)

Exclusion Criteria:

* Known hypersensitivity to fucoidan or seaweed products
* Currently using any other pharmacologic agents to specifically treat fatigue including psychostimulants or antidepressants. Note: Antidepressants used to treat items other than fatigue (such as hot flashes or depression) are allowed if the patient has been on a stable dose for ≥ 1 month prior to registration and plans to continue such for 8 weeks. Exercise is allowed
* Psychiatric disorder such as untreated/uncontrolled depression, manic depressive disorder, obsessive compulsive disorder or schizophrenia (defined per medical history)
* Surgery that required general anesthetic ≤ 4 weeks prior to registration
* Malnutrition, active infection, severe depression, significant pulmonary disease, and/or cardiovascular disease that the attending physician feels could be causing the patient's fatigue
* Use of any over-the-counter herbal/dietary supplement marketed for fatigue or energy (for example, products containing ginseng, rhodiola rosea, guarana, or anything called an "adaptogen"), including current use of fucoidan
* Current use of warfarin, heparin, enoxaparin, or a novel anticoagulant or known bleeding disorder/abnormal prothrombin time (PT)/partial thromboplastin time (PTT) at baseline
* Current use of bevacizumab
* Untreated thyroid conditions
* Use of chemotherapy and/or immunotherapy ≤ 90 days prior to registration
* Unwillingness to follow study related procedures
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue, weeks 1-8 | Baseline to 8 weeks
  Will be assessed using self-reported fatigue over the past week. Fatigue is rated on a scale of 0-10 where 0=no fatigue at all and 10=fatigue as bad as it can be. Fatigue scores will be compared between arms.

SECONDARY OUTCOMES:
Change in fatigue, weeks 9-16 | Baseline to 16 weeks
  Will be assessed using self-reported fatigue over the past week. Fatigue is rated on a scale of 0-10 where 0=no fatigue at all and 10=fatigue as bad as it can be. Fatigue scores will be compared between arms.
Change in the symptoms | Baseline to 16 weeks
  Will be measured using the Functional Assessment of Cancer Therapy-Fatigue (FACT-F) scores, a 13-item questionnaire assessing fatigue symptoms over the past week. Responses to each item are scored on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Scores will be compared between arms.
Change in Subjective Global Impression of Change scores | Week 8 and Week 16
  Will be measured using the Subjective Global Impression of Change instrument, which consists of 3 items assessed since beginning study medication: fatigue, emotional state, and overall quality of life. Items are scored on a 7-poin scale ranging from -3 (very much worse) to 3 (very much better). Two additional questions are answered only at the end of week 8: which medication the respondent believes they were on (2 choices) and whether they were satisfied with the effect of treatment on fatigue (yes/no).
Incidence of rates of symptoms | Up to 16 weeks
  Symptoms will be reported by the patient using the Symptom Experience Diary, which consists of 7 items assessing specific symptoms over the past week. Items are answered on a scale of 0 (none at all) to 10 (as bad as it can be). There is also one yes/no question related to exercise and one question for any side effects not addressed in the initial 7 items. Responses will be compared between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Zoey I. Harris, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials